CLINICAL TRIAL: NCT03912025
Title: The Relationship Between Having a Positive Mindset and Exercise Capacity in Patients With Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Naomi Gauthier, Pediatric Cardiologist, Boston Children's Hospital
Other Study IDs: P00030619
Record Dates: First submitted 2019-04-10; First posted 2019-04-11 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-04

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mild hemodynamic CHD: "Mild" severity category will be defined in terms of hemodynamic parameters rather than anatomic diagnoses, as outlined in the European Society of Cardiology Section on Sports Cardiology consensus guidelines (Budts W, Borjesson M, Chessa M, van Buuren F, Trindade PT, Corrado D, Heidbuchel H, Web G, Holm J, Papadakis M. 2013).
  They define functional parameters such as systolic function, oxygen saturation, rhythm disorders, elevated pressure or volume load, etc. to divide patients into 3 hemodynamic groups. Based on their model, we define "mild CHD" as ones falling into the group that can train at "High Intensity" exercise levels.
  Interventions: Other: Relationship between positive mindset and exercise capacity
- Moderate hemodynamic CHD: "Moderate" severity category will be defined in terms of hemodynamic parameters rather than anatomic diagnoses. Based on their model, we define "moderate CHD" as those that can train at "Moderate Intensity."
  Interventions: Other: Relationship between positive mindset and exercise capacity

INTERVENTIONS:
Other: Relationship between positive mindset and exercise capacity — No intervention. Cross-sectional study looking at the relationships between questionnaire scores and outcomes

SUMMARY:
A cross sectional study utilizing congenital heart disease patients presenting for clinically indicated cardiopulmonary exercise test. Baseline questionnaires (see below) will be administered prior to the exercise test. Exercise test data and clinical data will be recorded. Questionnaire data will be compared to clinical data in and between disease severity groups. Disease severity will be determined based on hemodynamic (not anatomic) classification according to an algorithm adapted from the European Society of Cardiology.

DETAILED DESCRIPTION:
Patients with congenital heart disease (CHD) have variable degrees of exercise capacity and levels of physical activity that is not necessarily related to disease severity (1,2) and is not fixed as supervised exercise training can achieve improved fitness across a spectrum of hemodynamic deficits (3-5). Effectiveness of training relates to frequency, intensity, time, and type of exercise as well as motivation to participate. Research in the psychology literature in athletes and in non-athletes alike has demonstrated that optimism and positive mentality result in improved exercise capacity, enhanced training results, and resilience to stress (6-11). Further, the general concept of resilience in children may be the sum result of the balance of positive and negative inputs (12), and these factors are also modifiable. The degree with which having a positive mindset impacts functional capacity irrespective of congenital heart disease severity is not known; if there is a correlation, then the idea that mindset could potentially be a target for an intervention to improve health in children with CHD is intriguing.

This study seeks to assess the correlation of positive thinking to physiological outcomes by comparing the degree of positive mindset of patients with congenital heart disease (as measured by questionnaire data to assess the balance of optimistic thinking to anxiety) with their functional capacity (as measured by peak oxygen consumption (peakVO2) on exercise testing). The ability to measure "mindset" in the clinic setting is now feasible after the recent release of a set of validated questionnaires for children (and parent-proxies) known as PROMIS (Patient-Reported Outcomes Measurement Information System), developed under the auspices of the National Institutes of Health (www.healthmeasures.net/explore-measurement-systems/promis). These questionnaires are short (4-8 questions), free, and integrate into the Research Electronic Data Capture (REDCap) database, making delivery Health Insurance Portability and Accountability Act (HIPAA) compliant and scoring automatic. In addition, the PROMIS measures contain both retrospective positive quality of life questions (life satisfaction, positive well-being) as well as a future facing tool measuring degree of optimism and purpose, making it ideally suited for the present research proposal. While PROMIS tools have been utilized in childhood chronic illnesses such as arthritis and kidney disease, they have not yet been reported in children with congenital heart disease. Thus, a secondary goal of this proposal is to assess the distribution of meaning and purpose scores and anxiety scores of children with CHD compared to the population norms.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 8-17 with congenital heart disease
* Classified as mild or moderate hemodynamic severity
* Presenting to outpatient department for clinically indicated cardiopulmonary exercise test

Exclusion Criteria:

* Patients on beta blockers or negative inotropes
* Patients with pacemakers/ICDs
* Patients with active arrhythmias
* Patients with significant musculoskeletal or pulmonary disease
* Patients unable to complete a maximal exercise test or for whom an exercise test is contraindicated
* Patients who are not fluent in English
* Patients unable to complete the questionnaire
* Patients who have severely hemodynamic debilitation or at risk (severe systolic dysfunction, severe ventricular hypertrophy, severe pressure load, severe volume load, severe pulmonary hypertension, malignant arrhythmia, significant central cyanosis)

Ages: 8 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Congenital Heart disease Patients
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-25 (Actual)

PRIMARY OUTCOMES:
Patient Reported Outcomes Measurement Information System (PROMIS) Pediatric Meaning and Purpose Score | up to 60 minutes
  A series of 8 questions that ask about future hopes, created and validated by a branch of the National Institutes of Health (www.healthmeasures.net). The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured. For positively-worded concepts like Meaning and Purpose, a T-score of 60 is one SD better than average. By comparison, a Meaning and Purpose T-score of 40 is one SD worse than average.
Patient Reported Outcomes Measurement Information System Pediatric Anxiety Score | up to 60 minutes
  A series of 8 questions to assess the degree of anxiety felt in the past week, created and validated by a branch of the National Institutes of Health (www.healthmeasures.net). The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation (SD) of 10. For negatively-worded concepts like anxiety, a T-score of 60 is one SD worse than average. By comparison, an anxiety T-score of 40 is one SD better than average.
Ratio of Meaning and Purpose Score to Anxiety Score | up to 60 minutes
  Since positive mindset is represented by a high score on the Meaning and Purpose scale, and a low score on the Anxiety scale, patients with high ratios (greater than 1) will have the most positive mindsets, while those with low ratios (less than 1) will have the least positive mindsets.

SECONDARY OUTCOMES:
Patient Reported Outcomes Measurement Information System Physical Activity Questionnaire | up to 60 minutes
  Self-reported physical activity questionnaire, created and validated by a branch of the National Institutes of Health (www.healthmeasures.net). The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation (SD) of 10. For positively-worded concepts like Physical Activity, a T-score of 60 is one SD better than average. By comparison, a Physical Activity T-score of 40 is one SD worse than average.
Patient Reported Outcomes Measurement Information System Pediatric Life Satisfaction Score | up to 60 minutes
  A series of 8 questions used as markers of current and recent (but not future) positive functioning, created and validated by a branch of the National Institutes of Health (www.healthmeasures.net). The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation (SD) of 10. For positively-worded concepts like Life Satisfaction, a T-score of 60 is one SD better than average. By comparison, a Life Satisfaction T-score of 40 is one SD worse than average.
Patient Reported Outcomes Measurement Information System Pediatric Positive Affect/Well Being Score | up to 60 minutes
  A series of 8 questions assessing friendships, created and validated by a branch of the National Institutes of Health (www.healthmeasures.net). The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation (SD) of 10. For positively-worded concepts like Positive Affect, a T-score of 60 is one SD better than average. By comparison, a Positive Affect T-score of 40 is one SD worse than average.
Pediatric Cardiac Quality of Life Inventory Questionnaire (PCQLI) | up to 60 minutes
  A standard quality of life tool for congenital heart disease. Three scores are generated: Disease Impact subscale score, Psychosocial Impact subscale score, and Total score. Disease Impact subscale score (up to 50 points) + Psychosocial Impact subscale score (up to 50 points) = Total score, for a maximum of 100 points. Higher scores represent better perceived health related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Gauthier, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No